CLINICAL TRIAL: NCT04424810
Title: Effect of High-quality Pre-operative Videos on Patient Anxiety Levels Prior to Ambulatory Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Christopher Larsen, Physician, Department of Orthopaedic Surgery, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0516
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Anxiety; Carpal Tunnel Syndrome; Trigger Finger; Engagement, Patient; Pain
MeSH Terms: conditions — Anxiety Disorders; Carpal Tunnel Syndrome; Trigger Finger Disorder; Patient Participation; Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel, 2 groups, 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Patients selected to be in the intervention group will be asked to watch a high-quality, physician created video describing their condition and the operative treatment they are about to undergo.
  Interventions: Other: High-quality, physician created video
- Control group (Placebo Comparator): Patients selected to be in the control group will not be asked to watch a video prior to surgery.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: High-quality, physician created video — The intervention group will watch a short (2-5 minute) video prior to surgery that will provide them with information about their condition and the procedure they are about to undergo (either carpal tunnel release or trigger finger release).
  Arms: Video group
Other: Standard of care — Patients in the control group will not be asked to do anything differently prior to their surgery
  Arms: Control group

SUMMARY:
Previous research has shown that YouTube is a poor source of high-quality medical information. This is likely because there is no regulation of the content on YouTube and relatively little of the content is posted by qualified medical professionals. It is known that up to 30% of patients use the internet to research the procedure they will be having and given the increasing popularity of YouTube we suspect many patients are using YouTube or similar sites as a source of information prior to elective surgery. There are likely a number of patient factors that contribute to patients seeking out videos as a source of pre-operative medical information. Patient age, which is generally inversely correlated to computer literacy, may have a role. Patient anxiety and pre-operative worrying may cause a patient to turn to the internet to search for information, and the poor overall quality of the content available may worsen pre-operative anxiety.

The primary objective of this study is to determine if providing patients with a reliable, high-quality video about their condition and operation prior to surgery reduces pre-operative anxiety. Secondary aims are to determine the percentage of patients that independently seek out videos online as a source of medical information prior to elective hand surgery, identify patient attributes that are associated with this behavior, and understand if introducing high quality pre-surgical videos has an impact on post-operative patient outcomes and/or patient engagement. The investigators hypothesize that providing patients with high-quality pre-operative videos will reduce pre-operative anxiety. Its is also expected that patients who seek out videos on their own for pre-operative medical information will be younger and have higher anxiety levels and pain catastrophizing scores. Additionally, the investigators hypothesize that patients who watch high-quality pre-operative videos may have better short term post-operative outcomes and greater engagement in their care than their counterparts that did not watch videos or who sought out videos on their own.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a primary routine elective hand procedure (Carpal tunnel release, trigger finger release)
* age > 18 years

Exclusion Criteria:

* revision procedure
* prior debilitating upper extremity injury
* surgery not being performed on ambulatory basis
* special populations (pregnant patients, prisoners or other institutionalized patients, cognitive impairment)
* non-english speaking patients (videos only available in english language)
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Pre-operative anxiety | Immediately prior to surgery
  We will measure pre-operative anxiety using the State-Trait Anxiety Inventory (STAI) 6-item short form (minimum score: 20, maximum score: 80, higher scores indicate more anxiety)

SECONDARY OUTCOMES:
Percentage of patients who sought out pre-operative videos before surgery | Immediately before surgery
  We plan to determine the percentage of patients who sought out pre-operative videos before surgery on websites such as YouTube as a part of our "video questionnaire"
Pain catastrophizing | Immediately before surgery
  As determined by the pain catastrophizing scale (PCS); (minimum score: 0, maximum score: 100, higher scores indicate more anxiety)
Patient engagement | Immediately before surgery
  To determine patient levels of engagement in their care as assessed by the Patient Activation Measure (PAM)-13 (minimum score: 0, maximum score: 100, higher scores indicate higher levels of activation/engagement in care)
Pain scores | At 48-72 hour post-operatively and 2 weeks post-operatively
  Assessed by Visual Analog Scale (VAS) pain scores (minimum: 0, maximum: 10, higher scores indicate greater levels of pain)
Functional outcomes | At 48-72 hour post-operatively and 2 weeks post-operatively
  Assessed by the Quick Disabilities of the Arm, Shoulder and Hand (qDASH) questionnaire (minimum: 0, maximum: 100, greater scores indicate a greater level of disability)

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Schwartz Ambulatory Surgery Center, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No